CLINICAL TRIAL: NCT01384799
Title: A Phase I Dose Escalation Study to Investigate the Safety and Pharmacokinetics of Intravenous CUDC-101 With Concurrent Cisplatin and Radiation Therapy in Subjects With Locally Advanced Head and Neck Cancer
Brief Title: Phase I Study of CUDC-101 With Cisplatin and Radiation in Subjects With Head & Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUDC-101-103
Record Dates: First submitted 2011-06-17; First posted 2011-06-29 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — 7-(4-(3-ethynylphenylamino)-7-methoxyquinazolin-6-yloxy)-N-hydroxyheptanamide; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CUDC-101 — CUDC-101 will be administered as a 1 hour intravenous infusion three times per week for a one week run-in (week -1) and then as part of the combination treatment on weeks 1-7. If the 225 mg/m2 dose is tolerated in the first cohort, the dose will be increased to 275 mg/m2. If the 225 mg/m2 dose is not tolerated, the dose will be decreased to 175 mg/m2. If 175 mg/m2 is not tolerated the dose will be further decreased to 150 mg/m2.
Drug: Cisplatin — Cisplatin will be administered intravenously at a dose of 100 mg/m2 on days 2, 23 and 44 of the seven week combination treatment course.
  Other Names: cisplatinum; CDDP; Platinol
Radiation: Radiation Therapy — The initial target volume encompassing the gross and subclinical disease sites will receive 2.0 Gy per fraction, five fractions per week. The gross disease sites will receive 70 Gy in 35 fractions over seven weeks and the subclinical disease sites will receive 56 Gy in 35 fractions, again over seven weeks.

SUMMARY:
This is a phase I dose escalation study of CUDC-101 in combination with concurrent cisplatin and radiation therapy in patients with locally advanced head and neck cancer. CUDC-101 is a multi-targeted agent designed to inhibit epidermal growth factor receptor (EGFR), human epidermal growth factor receptor Type 2 (Her2) and histone deacetylase (HDAC). The study is designed to establish the safety, tolerability and maximum tolerated dose (MTD) of CUDC-101 when administered in combination with concurrent cisplatin and radiation over an 8-week treatment course, consisting of a one week run-in period of CUDC-101 administered alone, followed by seven weeks of combination treatment with CUDC-101, cisplatin and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with locally advanced, pathologically confirmed diagnosis of squamous cell carcinoma of the head and neck at the following sites: oral cavity, oropharynx, hypopharynx and larynx with either:

  * Stage IV p16 positive tumors and >10 pack-years smoking history.
  * Stage III/IV p16 negative tumors, regardless of smoking history.
* At least evaluable disease; one measurable site of disease according to RECIST (Version 1.1) criteria (at least 10 mm for conventional CT/MRI or spiral CT scan) is desirable.
* Subjects enrolled in the MTD expansion cohort must have at least 1 tumor lesion that is suitable for repeat biopsy (pre- and post-CUDC-101 infusion).
* Age ≥ 18 years
* ECOG performance < 2
* Life expectancy ≥ 3 months
* If female, neither pregnant nor lactating
* If of child bearing potential, must use adequate birth control throughout the participation in the treatment phase and for 60 days following the last study treatment.
* Absolute neutrophil count ≥ 1,800/µL; platelets ≥ 100,000/µL; hemoglobin ≥ 8.0 g/dL, creatinine ≤ 1.5x upper limit of normal (ULN); total bilirubin ≤ 1.5x ULN; AST/ALT ≤ 2 x ULN.
* Serum magnesium and potassium within normal limits (may be supplemented to achieve normal values)
* Able to render informed consent and to follow protocol requirements.

Exclusion Criteria:

* Prior radiotherapy to the region of the study cancer or adjacent anatomical sites, or > 25% of marrow-bearing area.
* Prior chemotherapy for the current indication.
* Prior therapy that specifically and directly targets EGFR, HER2 or HDAC.
* Use of investigational agent(s) within 30 days prior to study treatment.
* Primary tumor site of nasopharynx, sinuses, or salivary gland.
* History of cardiac disease with a New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF), myocardial infarction (MI) or unstable angina in the past 6 months prior to Day 1 of treatment, serious arrhythmias requiring medication for treatment.
* Patients with prolonged QTc Interval >450 msec.
* Acquired Immune Deficiency Syndrome (AIDS) or known infection with human immunodeficiency virus (HIV). Testing is not required.
* Known history of gastrointestinal bleeding, ulceration, or perforation within 6 months prior to study treatment.
* Known history of stroke or cerebrovascular accident within 6 months prior to study treatment.
* Symptomatic cardiac conduction abnormality within 12 months prior to study treatment.
* Prior history of hearing impairment.
* Known history of renal disease or ongoing renal impairment.
* Any uncontrolled condition (such as active systemic infection, diabetes, hypertension), which in the opinion of the investigator, could affect the subjects participation in the study.
* Prior allergic reaction to cisplatin, carboplatin or other platinum-containing compounds.
* Central nervous system metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The number of participants with adverse events. | 18-24 months
  Safety and tolerability will be assessed by evaluating the number of patients with adverse events

SECONDARY OUTCOMES:
The number of subjects disease free at the completion of the treatment period. | 18-24 months
  To evaluate the efficacy of CUDC-101 in combination with cisplatin and radiation therapy by evaluating the number of subjects disease free at the completion of the treatment period.
The number of subjects disease free in the follow up period. | 18-24 months
  To evaluate the efficacy of CUDC-101 in combination with cisplatin and radiation therapy by evaluating the number of subjects disease free in the follow up period.
Concentration of CUDC-101 in the blood over time. | 18-24 months
  Pharmacokinetics will involve a determination of the concentration of CUDC-101 in the blood over time.
Number of circulating tumor cells pre treatment on Day -7 and 1 hour post treatment on Day -3. | 18-24 months
  The ability of CUDC-101 to exert a biological effect on the tumor will be examined in pharmacodynamic samples.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Overton Brooks VA Medical Center, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee